CLINICAL TRIAL: NCT04849507
Title: BabyStrong taVNS-Paired Bottle Feeding to Improve Oral Feeding
Brief Title: BabyStrong Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) Paired Bottle Feeding to Improve Oral Feeding
Acronym: BabyStrong I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 108881; 1R41HD104409 (NIH)
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Infant Feeding Problems, taVNS

STUDY DESIGN:
Intervention Model Description: If progress in daily oral feeding volumes is <4ml/kg/d after 10 days with either treatment A or B, we will offer cross-over to the alternate treatment, remaining blinded to treatment assignment.
Who Masked: Participant, Outcomes Assessor
Masking Description: blinded to study treatment assignment to active or sham taVNS. Perceptual threshold (PT) will be determined in both treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- active taVNS cymba to tragus (Active Comparator): We will deliver taVNS with the ear electrode positioned on left cymba and tragus, with pulses paired with oral feeding, off with rest during 2 feeds a day. Current will be delivered at 0.1milliAmpere (mA) < perceptual threshold (PT), 500microseconds, 25 Hertz (Hz).The ear electrode will be positioned on left tragus for active taVNS.
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- sham taVNS cymba to tragus (Sham Comparator): The ear electrode positioned on left cymba and tragus and as for active taVNS. We will test the PT with active stimulation, and then program a sham setting on the BabyStrong unit to deliver no current after the PT is determined.
  Interventions: Device: Sham transcutaneous auricular vagus nerve stimulation
- active taVNS cymba to mastoid (Active Comparator): We will deliver taVNS with the ear electrode positioned on left cymba and mastoid, with pulses paired with oral feeding, off with rest during 2 feeds a day. Current will be delivered at 0.1milliAmpere (mA) < perceptual threshold (PT), 500microseconds, 25 Hertz (Hz).The ear electrode will be positioned on left tragus for active taVNS.
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- sham taVNS cymba to mastoid (Sham Comparator): The ear electrode positioned on left cymba and mastoid as for active taVNS. We will test the PT with active stimulation, and then program a sham setting on the BabyStrong unit to deliver no current after the PT is determined.
  Interventions: Device: Sham transcutaneous auricular vagus nerve stimulation
- active taVNS cross over to sham (Experimental): infants who received 10 days of active taVNS but had <4ml/kg/d of oral feeding increase and crossed over the alternative treatment of sham taVNS
  Interventions: Device: transcutaneous auricular vagus nerve stimulation; Device: Sham transcutaneous auricular vagus nerve stimulation
- sham taVNS cross over to active taVNS (Experimental): infants who received 10 days of sham taVNS and had <4ml/kg/d of oral feeding increase and crossed over the alternative treatment of active taVNS
  Interventions: Device: transcutaneous auricular vagus nerve stimulation; Device: Sham transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
  Other Names: active taVNS
  Arms: active taVNS cross over to sham; active taVNS cymba to mastoid; active taVNS cymba to tragus; sham taVNS cross over to active taVNS
Device: Sham transcutaneous auricular vagus nerve stimulation — Sham stimulation of the left auricular branch of the vagus nerves paired with oral feeding
  Other Names: sham taVNS
  Arms: active taVNS cross over to sham; sham taVNS cross over to active taVNS; sham taVNS cymba to mastoid; sham taVNS cymba to tragus

SUMMARY:
Feeding is critical for pre-term infants and term infants with hypoxic ischemic brain injury, in order to be discharged home with their families and avoid a gastrostomy tube (G-tube) placement. The proposed study will employ a novel system that stimulates the vagus nerve through the skin in front part of the ear, the BabyStrong feeding system, to delivered transcutaneous auricular vagus nerve stimulation (taVNS) paired with oral feedings daily for 10 days. In an earlier study at Medical University of South Carolina (MUSC), this type of vagus nerve stimulation resulted in more than half of infants who were slated to receive G-tubes, taking full oral feeds by mouth and avoiding a G-tube. In this study some babies will receive the therapy for 10 days and others will get no stimulation. If no progress is made in feeding volumes by day 10, the infants will be switched to the other treatment for 7 days. Parents, study personnel, and care providers will be blinded to taVNS assignment. The electronic stimulation device is Federal Drug Administration (FDA)-cleared for investigational use, and the BabyStrong has been designated a Breakthrough Medical Device by the FDA. This study will be conducted in MUSC's Neonatal Intensive Care Unit.

DETAILED DESCRIPTION:
In this Phase I study, we will conduct a small-scale safety and feasibility study of 2 different taVNS units and ear electrode positions to optimize the BabyStrong portable taVNS feeding system and test the study design of randomization for 10 days. We will test the BabyStrong feeding system using up to n=10 active and n=10 sham taVNS in infants with twice daily treatment for 10 days, with cross over to alternate treatment for another 7days if there is no progress with feeds (increase <4ml/kg/d). G-tube placement will be arranged if infant continues to make no progress. If the infant attains full oral feeds and gains weight, they may be discharged at any time during the treatment protocol. The treatment assignment will be blinded to care providers, study personnel and parents. We will compare the number of participants who attain full oral feeds (= or > 130ml/kg/d with weight gain). Safety measures will be bradycardia and discomfort.

Criteria for success of BabyStrong feeding system: No sustained increase in discomfort scores; No bradycardia; attainment of full oral feeds in 50% of infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at any gestational age (GA), failing oral feeds after trying to learn feeding for 2 weeks if term, and 4 weeks if preterm
* safe to attempt oral feeds every feed without volume limitations by occupational or speech therapists, and
* clinical team is considering the need for a G-tube.

Exclusion Criteria:

* cardiomyopathy
* unstable bradycardia
* significant respiratory support
* infants of poorly controlled diabetic mothers, defined by obstetrical care providers, HgbA1C>5.6% or ketonuria.

Ages: 2 Weeks to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share our extensive database generated during the conduct of this study with other interested researchers on a collaborative basis, including developmental assessment and neuroimaging data associated with this study. Data will be de-identified consistent with Institutional Review Board (IRB) regulations and approval, as well as NIH data sharing policies.
Supporting Information: Study Protocol
Time Frame: after primary data analysis is complete, pending FDA review
Access Criteria: We will identify where the data will be available and how to access the data in any publications and presentations that we author or co-author about these data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment in the neonatal intensive care unit MUSC from 8/1/22 to 5/30/24
Pre-assignment Details: n=1 participant made rapid advance in feeds during screening studies prior to receiving any assigned treatment; Design includes a cross-over to alternative blinded treatment if feeding volume increase was <4ml/kg/d
  *participants only cross over between Active and Sham treatments within the same location
Groups:
- active taVNS unit tragus/ cymba conchae: We will deliver taVNS via the taVNS unit with the ear electrode positioned on left tragus or at the cymba conchae with return to the tragus. Pulses are paired with oral feeding, off with rest during 2 feeds a day. Current will be delivered at 0.1milliAmpere (mA) < perceptual threshold (PT), 500microseconds, 25 Hertz (Hz).
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- sham taVNS unit tragus/cymbae conchae: We will deliver inactive /sham taVNS via the taVNS unit with the ear electrode positioned around left cymba conchae/ inner tragus with return to the outer tragus. No pulses are delivered when pressing trigger, paired with oral feeding during 2 feeds a day. No current will be delivered, and assignment will be blinded.
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- Active taVNS unit cymba conchae/mastoid: We will deliver taVNS via the taVNS unit on the vagus channel with the ear electrode positioned around left cymba conchae with return to the mastoid. Pulses are paired with oral feeding, off with rest during 2 feeds a day. Current will be delivered at 0.1milliAmpere (mA) < perceptual threshold (PT), 500microseconds, 25 Hertz (Hz).
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- Sham taVNS unit cymbae conchae/mastoid: We will deliver inactive /sham taVNS via the aVNS unit on the vagus channel with the ear electrode positioned around left cymba conchae with return to the mastoid. No pulses are delivered when pressing trigger, paired with oral feeding during 2 feeds a day. No current will be delivered, and assignment will be blinded.
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- Active taVNs crossover to sham taVNS: infants who received 10 days of active taVNS but had <4ml/kg/d of oral feeding increase and crossed over the alternative treatment of sham taVNS
Period: Overall Study
Arm/Group | active taVNS unit tragus/ cymba conchae | sham taVNS unit tragus/cymbae conchae | Active taVNS unit cymba conchae/mastoid | Sham taVNS unit cymbae conchae/mastoid | Active taVNs crossover to sham taVNS | Sham taVNS cross over to active taVNS
Started | 5 | 3 | 2 | 2 | 2 | 2
cross over to alternate treatment (crossover to alternative treatment if oral feeding volume was increasing by < 4ml/kg/d) | 0 | 0 | 0 | 0 | 2 | 2
Completed | 5 | 3 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham taVNS unit cymbae conchae/mastoid: We will deliver inactive /sham taVNS via the taVNS unit on the vagus channel with the ear electrode positioned around left cymba conchae with return to the mastoid. No pulses are delivered when pressing trigger, paired with oral feeding during 2 feeds a day. No current will be delivered, and assignment will be blinded.
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- active taVNS crossover to sham taVNS: We deliver taVNS via the taVNS unit with the ear electrode positioned on left tragus or at the cymba conchae with return to the tragus. Pulses are paired with oral feeding, off with rest during 2 feeds a day. Current will be delivered at 0.1milliAmpere (mA) < perceptual threshold (PT), 500microseconds, 25 Hertz (Hz). Following 10 days of active stimulation with feeds, if infant is making < 4ml/kg/day increase in oral feed volume we will cross over to sham taVNS for up to 7 days of twice daily treatment.
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- Sham taVNS cross over to active taVNS: We deliver taVNS via the taVNS unit with the ear electrode positioned on left tragus or at the cymba conchae with return to the tragus. No active pulses are paired with oral feeding, for the sham condition during 2 feeds a day. Following 10 days of sham stimulation with feeds, if infant is making < 4ml/kg/day increase in oral feed volume we will cross over to active taVNS for up to 7 days of twice daily treatment with current will be delivered at 0.1milliAmpere (mA) < perceptual threshold (PT), 500microseconds, 25 Hertz (Hz).
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- Total: Total of all reporting groups
Arm/Group | active taVNS unit tragus/ cymba conchae | sham taVNS unit tragus/cymbae conchae | Active taVNS unit cymba conchae/mastoid | Sham taVNS unit cymbae conchae/mastoid | active taVNS crossover to sham taVNS | Sham taVNS cross over to active taVNS | Total
Number analyzed (Participants) | 5 | 3 | 2 | 2 | 2 | 2 | 16
Age, Continuous [Mean (Full Range); unit: weeks] — post menstrual age
  weeks | 41.2 [39.3 to 43.5] | 44.6 [40.3 to 50.9] | 42.8 [41.5 to 44] | 43.6 [43.6 to 43.7] | 48.6 [41.9 to 55.4] | 41.5 [40.5 to 42.4] | 43.5 [39.3 to 55.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 1 | 2 | 0 | 8
  Male | 2 | 2 | 1 | 1 | 0 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 2 | 2 | 2 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 1 | 1 | 1 | 7
  White | 2 | 1 | 2 | 0 | 1 | 1 | 7
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bradycardia
Description: safety : number of participants with episode of Heart rate < 80beats per minute for 5 seconds, according to the first assigned treatment
Time Frame: 30 minutes during taVNS paired-feed for 10 days
Population: Crossover arms are exploratory due to the small sample size.
Measure: Count of Participants; unit: Participants
Groups:
- active taVNS cross over to sham taVNS: Infants who receive 10 days of active taVNS twice daily with feeds, but have <4ml/kg/d increase in daily oral feed volume and cross over to alternative treatment of sham taVNS for up to 7 days
- Sham taVNS cross over to active taVNS: Infants who receive 10 days of sham taVNS twice daily with feeds, but have <4ml/kg/d increase in daily oral feed volume and cross over to alternative treatment of active taVNS for up to 7 days
Arm/Group | active taVNS unit tragus/ cymba conchae | sham taVNS unit tragus/cymbae conchae | Active taVNS unit cymba conchae/mastoid | Sham taVNS unit cymbae conchae/mastoid | active taVNS cross over to sham taVNS | Sham taVNS cross over to active taVNS
Number analyzed (Participants) | 5 | 3 | 2 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Discomfort Scores
Description: mean number of participants with Neonatal and Infant Pain scale (NIPS) >3 point increase, indicating worse discomfort according to the first assigned treatment
Time Frame: 30 minutes during taVNS paired-feed up to 17 days
Population: Crossover arms are exploratory due to the small sample size.
Measure: Count of Participants; unit: Participants
Arm/Group | active taVNS unit tragus/ cymba conchae | sham taVNS unit tragus/cymbae conchae | Active taVNS unit cymba conchae/mastoid | Sham taVNS unit cymbae conchae/mastoid | active taVNS cross over to sham taVNS | sham taVNS cross over to active taVNS
Number analyzed (Participants) | 5 | 3 | 2 | 2 | 2 | 2
Participants | 1 | 3 | 1 | 0 | 0 | 0

3. Primary Outcome: Participants Who Attain Full Oral Feeds
Description: taVNS in participants who received tragus stimulation and attained full oral feeds (oral intake = or >130ml/kg/day with weight gain) according to the first assigned treatment
Time Frame: 17 days
Population: Crossover arms are exploratory due to the small sample size.
Measure: Count of Participants; unit: Participants
Groups:
- Active taVNS cymba conchae to mastoid: We will deliver taVNS via the taVNS unit on the vagus channel with the ear electrode positioned around left cymba conchae with return to the mastoid. Pulses are paired with oral feeding, off with rest during 2 feeds a day. Current will be delivered at 0.1milliAmpere (mA) < perceptual threshold (PT), 500microseconds, 25 Hertz (Hz).
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- Sham taVNS cymba conchae to mastoid: We will deliver inactive /sham taVNS via the taVNS unit on the vagus channel with the ear electrode positioned around left cymba conchae with return to the mastoid. No pulses are delivered when pressing trigger, paired with oral feeding during 2 feeds a day. No current will be delivered, and assignment will be blinded.
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
Arm/Group | active taVNS unit tragus/ cymba conchae | sham taVNS unit tragus/cymbae conchae | Active taVNS cymba conchae to mastoid | Sham taVNS cymba conchae to mastoid | active taVNS cross over to sham taVNS | sham taVNS cross over to active taVNS
Number analyzed (Participants) | 5 | 3 | 2 | 2 | 2 | 2
Participants | 4 | 2 | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: collected over the acute treatment phase of the study (2-3 weeks) until Gastrostomy tube placement or discharge
Description: standard AE descriptions; Expected adverse events are reported as safety outcomes (Bradycardia, discomfort increase). there were no unanticipated AEs. limitations: initial treatment assignment may have an effect that cannot be washed-out by cross-over to the other treatment.
Groups:
- sham taVNS unit tragus/ cymba conchae: We will deliver inactive /sham taVNS via the taVNS unit with the ear electrode positioned around left cymba conchae/ inner tragus with return to the outer tragus. No pulses are delivered when pressing trigger, paired with oral feeding during 2 feeds a day. No current will be delivered, and assignment will be blinded.
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- Sham taVNS unit cymba conchae/mastoid: We will deliver inactive /sham taVNS via the taVNS unit on the vagus channel with the ear electrode positioned around left cymba conchae with return to the mastoid. No pulses are delivered when pressing trigger, paired with oral feeding during 2 feeds a day. No current will be delivered, and assignment will be blinded.
  transcutaneous auricular vagus nerve stimulation: Stimulation of the auricular branch of the left vagus nerve paired with oromotor feeding.
- active taVNS crossover to sham taVNS: infants who received 10 days of active taVNS but had <4ml/kg/d of oral feeding increase and crossed over the alternative treatment of sham taVNS for up to 7 days
- sham taVNS cross over to active taVNS: infants who received 10 days of sham taVNS and had <4ml/kg/d of oral feeding increase and crossed over the alternative treatment of active taVNS for up to 7 days
Arm/Group | active taVNS unit tragus/ cymba conchae | sham taVNS unit tragus/ cymba conchae | Active taVNS unit cymba conchae/mastoid | Sham taVNS unit cymba conchae/mastoid | active taVNS crossover to sham taVNS | sham taVNS cross over to active taVNS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/2 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/2 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/2 | 0/2 | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
small phase I study not powered for statistical analysis; Expected adverse events are reported as safety outcomes (Bradycardia, discomfort increase). There were no unanticipated AEs. Limitations: initial treatment assignment may have an effect that cannot be washed-out by cross-over to the other treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT04849507/Prot_001.pdf
  • Informed Consent Form (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT04849507/ICF_000.pdf